CLINICAL TRIAL: NCT02513940
Title: Influence of Testosterone Administration on Drug-Induced QT Interval Prolongation and Torsades de Pointes
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Indiana University (Other)
Collaborators: American Heart Association (Other); Purdue University (Other)
Responsible Party: Principal Investigator, James E. Tisdale, Adjunct Professor, Indiana University
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Prevention
Other Study IDs: 1507526854
Record Dates: First submitted 2015-07-29; First posted 2015-08-03 (Estimated); Results first posted 2019-03-06 (Actual); Last update posted 2019-08-28 (Actual); Status verified 2019-08

CONDITIONS: Long QT Syndrome
Keywords: Torsades de pointes; Testosterone; Progesterone; Clinical trial; Risk reduction; Electrocardiography
MeSH Terms: conditions — Long QT Syndrome; Torsades de Pointes; Risk Reduction Behavior | interventions — Testosterone; Progesterone; Drugs, Generic; Lactose; ibutilide

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (6):
- Testosterone - progesterone - placebo (Experimental): Subjects received transdermal testosterone gel 1% 100 mg once daily in the morning and two (2) oral placebo capsules x 7 days. After a washout of at least 13 days, they then received oral progesterone 400 mg (2 x 200 mg capsules) once every evening for 7 days and transdermal placebo gel once daily every morning for 7 days. After a washout period of at least 13 days, they then received transdermal placebo gel once daily every morning for 7 days and oral placebo once daily every morning x 7 days
  Interventions: Drug: Testosterone; Drug: Progesterone; Drug: Placebo; Drug: Ibutilide
- Testosterone - placebo - progesterone (Experimental): Subjects received transdermal testosterone gel 1% 100 mg once daily in the morning and two (2) oral placebo capsules x 7 days. After a washout of at least 13 days, they then received transdermal placebo gel once daily every morning for 7 days and oral placebo ( 2 capsules) once daily every morning x 7 days. After a washout period of at least 13 days, they then received oral progesterone 400 mg (2 x 200 mg capsules) once every evening for 7 days and transdermal placebo gel once daily every morning for 7 days.
  Interventions: Drug: Testosterone; Drug: Progesterone; Drug: Placebo; Drug: Ibutilide
- Progesterone - testosterone - placebo (Experimental): Subjects received oral progesterone 400 mg (2 x 200 mg capsules) once every evening for 7 days and transdermal placebo gel once daily every morning for 7 days. After a washout period of at least 13 days, they then received transdermal testosterone gel 1% 100 mg once daily in the morning and two (2) oral placebo capsules x 7 days. After a washout period of at least 13 days, they then received transdermal placebo gel once daily every morning for 7 days and oral placebo (2 capsules) once daily every morning x 7 days
  Interventions: Drug: Testosterone; Drug: Progesterone; Drug: Placebo; Drug: Ibutilide
- Progesterone - placebo - testosterone (Experimental): Subjects received oral progesterone 400 mg (2 x 200 mg capsules) once every evening for 7 days and transdermal placebo gel once daily every morning for 7 days. After a washout period of at least 13 days, they then received transdermal placebo gel once daily every morning for 7 days and oral placebo (2 capsules) once daily every morning x 7 days. After a washout period of at least 13 days, they then received transdermal testosterone gel 1% 100 mg once daily in the morning and two (2) oral placebo capsules x 7 days.
  Interventions: Drug: Testosterone; Drug: Progesterone; Drug: Placebo; Drug: Ibutilide
- Placebo - testosterone - progesterone (Experimental): Subjects received transdermal placebo gel once daily every morning for 7 days and oral placebo once daily every morning x 7 days. After a washout period of at least 13 days, they then received transdermal testosterone gel 1% 100 mg once daily in the morning and two (2) oral placebo capsules x 7 days. After a washout period of at least 13 days, they then received oral progesterone 400 mg (2 x 200 mg capsules) once every evening for 7 days and transdermal placebo gel once daily every morning for 7 days.
  Interventions: Drug: Testosterone; Drug: Progesterone; Drug: Placebo; Drug: Ibutilide
- Placebo - progesterone - testosterone (Experimental): Subjects received transdermal placebo gel once daily every morning for 7 days and oral placebo once daily every morning x 7 days. After a washout period of at least 13 days, they then received oral progesterone 400 mg (2 x 200 mg capsules) once every evening for 7 days and transdermal placebo gel once daily every morning for 7 days. After a washout period of at least 13 days, they then received transdermal testosterone gel 1% 100 mg once daily in the morning and two (2) oral placebo capsules x 7 days.
  Interventions: Drug: Testosterone; Drug: Progesterone; Drug: Placebo; Drug: Ibutilide

INTERVENTIONS:
Drug: Testosterone — Subjects will receive transdermal testosterone gel 1% 100 mg daily for 7 days
  Other Names: Androgel
Drug: Progesterone — Subjects will receive oral progesterone 400 mg (two x 200 mg capsules) once daily every evening for 7 days
  Other Names: Generic
Drug: Placebo — Subjects will receive placebo transdermal gel and placebo (lactose) capsules
  Other Names: Lactose
Drug: Ibutilide — Ibutilide 0.003 mg/kg administered to all subjects in all phases to moderately lengthen the QT interval
  Other Names: Corvert

SUMMARY:
Torsades de pointes (TdP) is a potentially fatal ventricular arrhythmia associated with corrected QT (QTc) interval prolongation. More than 50 commonly used drugs available on the US market may cause QTc interval prolongation and TdP. While TdP occurs more commonly in women, 33-45% of all cases of TdP have occurred in men. Older age is a risk factor for drug-induced TdP in men, possibly due to declining serum testosterone concentrations. Available evidence shows an inverse relationship between QTc intervals and serum testosterone concentrations. In addition, experimental data, including those from the investigators' laboratory, suggest that both exogenous testosterone or progesterone administration may be protective against prolongation of ventricular repolarization and TdP. Specific Aim: Establish the influence of transdermal testosterone administration and oral progesterone administration as preventive methods by which to diminish the degree of drug-induced QT interval prolongation in men 65 years of age or older. Hypothesis: Transdermal testosterone administration and oral progesterone administration both effectively attenuate drug-induced QT interval response in older men. To test this hypothesis, transdermal testosterone, oral progesterone or placebo will be administered in a 3-way crossover study to men 65 years of age or older. QTc interval response to low-dose ibutilide will be assessed. The primary endpoints will be Fridericia-corrected QT interval (QTF) response to ibutilide, in the presence and absence of testosterone, and in the presence or absence of progesterone: 1) Effect on pre-ibutilide QTF, 2) Effect on maximum post-ibutilide QTF, 3) Effect on % change in post-ibutilide QTF, and 2) Area under the QTF interval-time curves.

ELIGIBILITY:
Inclusion Criteria:

* Men ≥ 65 years of age

Exclusion Criteria:

* Prostate cancer; history of prostate cancer;
* History of breast cancer; benign prostatic hypertrophy;
* Weight < 60 kg
* Weight > 135 kg
* Serum k+ < 3.6 mEq/L;
* Serum mg2+ < 1.8 mg/dL;
* Hemoglobin < 9.0 mg/dL;
* Hematocrit < 26%;
* Hepatic transaminases > 3x upper limit of normal;
* Baseline Bazett's-corrected QT interval > 450 ms
* Heart failure due to reduced ejection fraction (left ventricular ejection fraction < 40%)
* Family or personal history of long-QT syndrome, arrhythmias or sudden cardiac death;
* Concomitant use of any QT interval-prolonging drug.

Min Age: 65 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Older Adult
Enrollment: 14 (Actual)
Dates: Start 2016-05 (Actual); Primary Completion 2017-10-19 (Actual); Study Completion 2017-10-19 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: James E Tisdale, PharmD, Principal Investigator — Purdue University
Locations (1):
- Indiana University, Indianapolis, Indiana, United States

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Muensterman ET, Jaynes HA, Sowinski KM, Overholser BR, Shen C, Kovacs RJ, Tisdale JE. Effect of Transdermal Testosterone and Oral Progesterone on Drug-Induced QT Interval Lengthening in Older Men: A Randomized, Double-Blind, Placebo-Controlled Crossover-Design Study. Circulation. 2019 Sep 24;140(13):1127-1129. doi: 10.1161/CIRCULATIONAHA.119.041395. Epub 2019 Sep 23. No abstract available. PMID 31545681
- [Derived] Tomaselli Muensterman E, Jaynes HA, Sowinski KM, Overholser BR, Shen C, Kovacs RJ, Tisdale JE. Transdermal Testosterone Attenuates Drug-Induced Lengthening of Both Early and Late Ventricular Repolarization in Older Men. Clin Pharmacol Ther. 2021 Jun;109(6):1499-1504. doi: 10.1002/cpt.2072. Epub 2020 Nov 15. PMID 33020898

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Recruitment began in July 2015; procedures were completed on last enrolled subject in October 2017.
  Subjects were recruited from advertisements placed in a seniors magazine, assisted living facilities, and local health fairs.
Pre-assignment Details: n=77 subjects initially assessed for eligibility; n=16 declined to participate, n= 49 excluded (met one or more exclusion criteria); n=22 provided written informed consent (these participants were not considered to be enrolled); n= 8 excluded after providing consent because they were found to meet an exclusion criterion
Period: Overall Study
Arm/Group | Testosterone - Progesterone - Placebo | Testosterone - Placebo - Progesterone | Progesterone - Testosterone - Placebo | Progesterone - Placebo - Testosterone | Placebo - Testosterone - Progesterone | Placebo - Progesterone - Testosterone
Started | 2 (This was a crossover study, with a total n=14. All 14 subjects completed each phase of the study) | 3 | 2 | 2 | 2 | 3
Completed | 2 | 3 | 2 | 2 | 2 | 3
Not Completed | 0 | 0 | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Population: Men 65 years of age or older were enrolled
Groups:
- All Study Participants: Men 65 years of age or older were enrolled. Exclusion criteria were: prostate cancer; history of prostate or breast cancer; benign prostatic hyperplasia; weight < 60 kg or > 135 kg; serum potassium < 3.6 mEq/L; serum magnesium < 1.8 mg/dL; hematocrit < 26%; hepatic transaminases > 3x upper limit of normal; baseline Bazett's-corrected QTc interval > 450 ms; heart failure with reduced ejection fraction (left ventricular ejection fraction < 40%); family or personal history of long QT syndrome, arrhythmias or sudden cardiac death; permanently paced ventricular rhythm; concomitant use of any QT interval-prolonging drug or strong non-QT interval-prolonging cytochrome P450 3A inhibitors.
Arm/Group | All Study Participants
Number analyzed (Participants) | 14
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 1
  >=65 years | 13
Age, Continuous [Mean (Standard Deviation); unit: years] | 73 (6)
Age, Continuous [Mean (Standard Deviation); unit: Years] | 73 (6)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0
  Male | 14
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0
  Not Hispanic or Latino | 14
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 1
  White | 13
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  United States | 14
Weight [Mean (Standard Deviation); unit: kg] | 90 (16)

OUTCOME MEASURES:

1. Primary Outcome: Baseline (Pre-ibutilide) Individualized Rate-corrected QT Interval (QTF)
Description: QT interval is an electrocardiogram (ECG) measure of ventricular repolarization. Prolonged QT interval is a marker of increased risk of the ventricular arrhythmia known as torsades de pointes, which can cause sudden cardiac death. QT intervals were measured from ECG lead II by one investigator (E.T.M.) who was blinded to the subjects' assigned treatment phases. QT intervals were measured using computerized high-resolution electronic calipers (EP Calipers 1.6). QT and RR intervals at each time point were averaged over 3 consecutive complexes. The end of the T-wave was determined via the tangent method. Only clearly discernable QT intervals were measured. QT intervals vary with heart rate, and therefore must be corrected for heart rate. QT intervals were corrected using the Fridericia (QTF) method. The baseline QTF assesses the influence of testosterone and progesterone on naturally-occurring (before ibutilide administration) QTF
Time Frame: Following 7 days of testosterone, progesterone or placebo
Measure: Mean (Standard Deviation); unit: ms
Groups:
- Testosterone: Testosterone gel 1% 100 mg daily x 7 days
  Testosterone: Subjects will receive transdermal testosterone gel 1% 100 mg daily for 7 days
  Ibutilide: Ibutilide 0.003 mg/kg administered to all subjects in all phases to moderately lengthen the QT interval
- Progesterone: Progesterone 400 mg orally daily x 7 days
  Progesterone: Subjects will receive oral progesterone 400 mg (two x 200 mg capsules) once daily every evening for 7 days
  Ibutilide: Ibutilide 0.003 mg/kg administered to all subjects in all phases to moderately lengthen the QT interval
- Placebo: Dual matching placebo capsules and placebo topical gel every day x 7 days
  Placebo
  Ibutilide: Ibutilide 0.003 mg/kg administered to all subjects in all phases to moderately lengthen the QT interval
Arm/Group | Testosterone | Progesterone | Placebo
Number analyzed (Participants) | 14 | 14 | 14
ms | 393 (19) | 399 (16) | 399 (13)
Statistical Analysis 1: Comparison: Testosterone vs Progesterone vs Placebo; Test type: Superiority; p = 0.09, Mixed Models Analysis

2. Primary Outcome: Maximum QTF Following Ibutilide 0.003 mg/kg
Description: QT interval is an ECG measure of ventricular repolarization. Prolonged QT interval is a marker of increased risk of the ventricular arrhythmia known as torsades de pointes, which can cause sudden cardiac death. Three 12-lead ECGs were obtained ~ 1 minute apart immediately at the end of the ibutilide infusion and at 5, 10, 15, 20, 30, and 45 minutes and 1, 2, 4, 6, and 8 hours post-infusion. QT intervals were measured from ECG lead II by one investigator (E.T.M.) who was blinded to the subjects' assigned treatment phases. QT intervals were measured using computerized high-resolution electronic calipers. QT and RR intervals at each time point were averaged over 3 consecutive complexes. The end of the T-wave was determined via the tangent method. QT intervals vary with heart rate, and therefore must be corrected for heart rate. QT intervals were corrected using the Fridericia (QTF) method. Maximum QTF is the longest QTF measured following ibutilide at any time point.
Time Frame: Within 8 hours following ibutilide administration
Measure: Mean (Standard Deviation); unit: ms
Arm/Group | Testosterone | Progesterone | Placebo
Number analyzed (Participants) | 14 | 14 | 14
ms | 416 (19) | 425 (22) | 426 (18)
Statistical Analysis 1: Comparison: Testosterone vs Progesterone vs Placebo; Test type: Superiority; p = 0.001, Mixed Models Analysis — Pairwise comparisons: Testosterone vs placebo: p=0.008 Progesterone vs placebo: p=0.73 Testosterone vs progesterone: p=0.0008

3. Primary Outcome: Maximum Percent Change From Pretreatment Value in QTF Following Ibutilide 0.003 mg/kg
Description: QT interval is an ECG measure of ventricular repolarization. Prolonged QT interval is a marker of increased risk of the ventricular arrhythmia known as torsades de pointes, which can cause sudden cardiac death. Three 12-lead ECGs were obtained ~ 1 minute apart immediately at the end of the ibutilide infusion and at 5, 10, 15, 20, 30, and 45 minutes and 1, 2, 4, 6, and 8 hours post-infusion. QT intervals were measured from ECG lead II by one investigator (E.T.M.) who was blinded to the subjects' assigned treatment phases. QT intervals were measured using computerized high-resolution electronic calipers. QT and RR intervals at each time point were averaged over 3 consecutive complexes. The end of the T-wave was determined via the tangent method. QT intervals were corrected using the Fridericia (QTF) method.
Time Frame: Within 8 hours of ibutilide administration
Measure: Mean (Standard Deviation); unit: Percent change
Groups:
- Testosterone: Testosterone gel 1% 100 mg daily x 7 days Oral placebo capsules once daily for 7 days
  Testosterone: Subjects will receive transdermal testosterone gel 1% 100 mg daily for 7 days
  Ibutilide: Ibutilide 0.003 mg/kg administered to all subjects in all phases to moderately lengthen the QT interval
- Progesterone: Progesterone 400 mg orally daily x 7 days Transdermal placebo gel once daily for 7 days
  Progesterone: Subjects will receive oral progesterone 400 mg (two x 200 mg capsules) once daily every evening for 7 days
  Ibutilide: Ibutilide 0.003 mg/kg administered to all subjects in all phases to moderately lengthen the QT interval
Arm/Group | Testosterone | Progesterone | Placebo
Number analyzed (Participants) | 14 | 14 | 14
Percent change | 5.6 (1.8) | 5.9 (2.3) | 6.1 (1.9)
Statistical Analysis 1: Comparison: Testosterone vs Progesterone vs Placebo; Test type: Superiority; p = 0.60, Mixed Models Analysis; Repeated measures ANOVA

4. Secondary Outcome: Area Under the QTF Versus Time Curve for 0-1 Hour Following Ibutilide 0.003 mg/kg
Description: Prolonged QT interval is a marker of increased risk of the ventricular arrhythmia known as torsades de pointes, which can cause sudden cardiac death. Three 12-lead ECGs were obtained ~ 1 minute apart immediately at the end of the ibutilide infusion and at 5, 10, 15, 20, 30, and 45 minutes and 1, 2, 4, 6, and 8 hours post-infusion. QT intervals were measured from ECG lead II by one investigator (E.T.M.) who was blinded to the subjects' assigned treatment phases. QT intervals were measured using computerized high-resolution electronic calipers. QT and RR intervals at each time point were averaged over 3 consecutive complexes. The end of the T-wave was determined via the tangent method. Area under the QTF curve was calculated using the trapezoidal rule and reflects overall QTF interval "exposure" over time.
Time Frame: 1 hour following ibutilide administration
Measure: Mean (Standard Deviation); unit: ms·hr
Arm/Group | Testosterone | Progesterone | Placebo
Number analyzed (Participants) | 14 | 14 | 14
ms·hr | 471 (24) | 480 (24) | 483 (18)
Statistical Analysis 1: Comparison: Testosterone vs Progesterone vs Placebo; Test type: Superiority; p = 0.0003, Mixed Models Analysis — Pairwise comparisons: Testosterone vs placebo: p = 0.0001 Progesterone vs placebo: p = 0.25 Testosterone vs progesterone: p = 0.002; Repeated measures ANOVA

5. Secondary Outcome: Number of Participants With Adverse Effects Associated With Testosterone, Progesterone and Placebo
Description: Adverse effects were assessed by study investigators using telephone calls during the 7-day treatment period in each phase, as well as by asking participants about adverse effects on ibutilide administration days
Time Frame: During 7 day administration periods
Measure: Count of Participants; unit: Participants
Arm/Group | Testosterone | Progesterone | Placebo
Number analyzed (Participants) | 14 | 14 | 14
Participants
  Fatigue | 0 | 1 | 0
  Rash on gel application site | 0 | 0 | 1
Statistical Analysis 1: Comparison: Testosterone vs Progesterone vs Placebo; Fatigue; Test type: Superiority; p > 0.99, Fisher Exact
Statistical Analysis 2: Comparison: Testosterone vs Progesterone vs Placebo; Rash at gel application site; Test type: Superiority; p > 0.99, Fisher Exact

ADVERSE EVENTS:
Time Frame: 8 days per study phase
Arm/Group | Testosterone | Progesterone | Placebo
All-Cause Mortality (participants affected / at risk) | 0/14 | 0/14 | 0/14
Serious Adverse Events (participants affected / at risk) | 0/14 | 0/14 | 0/14
Other Adverse Events (participants affected / at risk) | 0/14 | 1/14 | 1/14
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Testosterone (N=14) | Progesterone (N=14) | Placebo (N=14)
Fatigue (General disorders) | 0 | 1 | 0
Rash on gel application site (Skin and subcutaneous tissue disorders) | 0 | 0 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2017-07-10): https://cdn.clinicaltrials.gov/large-docs/40/NCT02513940/Prot_SAP_001.pdf